CLINICAL TRIAL: NCT03893734
Title: Effect of Methadone and Hydromorphone on the QT Interval After Anesthesia and Surgery
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Endeavor Health (Other)
Responsible Party: Principal Investigator, Glenn Murphy, Director of Clinical Research, Endeavor Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: EH17-264
Record Dates: First submitted 2018-05-26; First posted 2019-03-28 (Actual); Last update posted 2019-09-13 (Actual); Status verified 2019-09

CONDITIONS: EKG-QT Prolongation
MeSH Terms: interventions — Methadone; Hydromorphone

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to receive either methadone at the start of anesthesia or hydromorphone at the end of surgery
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Clinicians will be provided with two blinded syringes containing either saline and hydromorphone or methadone and saline.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- methadone group (Active Comparator): Patients in this group will receive a syringe of methadone at the induction of anesthesia and a syringe of saline at the end of anesthesia.
  Interventions: Drug: methadone
- hydromorphone group (Placebo Comparator): Patients in this group will receive a syringe of saline at induction of anesthesia and a syringe of hydromorphone at the end of anesthesia
  Interventions: Drug: Hydromorphone

INTERVENTIONS:
Drug: methadone — Patients in the methadone group will receive a syringe of methadone at induction of anesthesia and a syringe of saline at the end of anesthesia
  Arms: methadone group
Drug: Hydromorphone — Patients in the hydromorphone group will receive a syringe of saline at induction of anesthesia and a syringe of hydromorphone at the end of anesthesia
  Arms: hydromorphone group

SUMMARY:
A number of drugs used in the perioperative period may cause prolongation of the QT interval on the electrocardiogram (EKG). These drugs include inhalational agents, antiemetic agents, pain medications, and drugs used to reverse the effects of muscle relaxants. Approximately 80% of patients undergoing a general anesthetic will demonstrate significant prolongation of the QT interval on the EKG in the postanesthesia care unit (PACU) following surgery. The concern with QT interval prolongation is that it can result in a potentially lethal ventricular arrhythmia termed torsade des pointes. Despite the concurrent use of several of these medications in a typical general anesthetic, torsade des pointes is a rare event in the perioperative period. In the past decade, the use of intravenous methadone as part of a balanced anesthetic technique has increased significantly. A single dose provided at induction of anesthesia can provide prolonged (24-48 hours) relief from pain. Studies in patients receiving long-term treatment with methadone for addiction therapy or chronic pain have revealed that these patients are at risk for QT prolongation, torsade des pointe, and cardiac death. However, the effect of a single intravenous dose of methadone used in the operating room on the QT interval is uncertain. The aim of this randomized clinical trial is to compare the impact of methadone, when compared to the more commonly-used opioid hydromorphone, on QT prolongation measured with a 12-lead EKG in the PACU and on postoperative day 1. We hypothesize that methadone will not result in significant QT prolongation when used as part of a standardized general anesthetic.

DETAILED DESCRIPTION:
In the past decade, the single most common cause of withdrawal of the use of drugs that have already been marketed has been the prolongation of the QT interval on the electrocardiogram associated with polymorphic ventricular tachycardia, or torsade de pointes. Without treatment, torsade de pointes can progress to a lethal ventricular arrhythmia. A number of drugs which prolong the QT interval can precipitate torsade de pointes. However, a number of risk factors are often present in patients who develop drug-induced torsade de pointes. These include hypomagnesemia, hypokalemia, female gender, bradycardia, congestive heart failure, rapid rate of drug infusion, and high drug concentrations. Exposure to a drug that prolongs the QT interval, particularly in a susceptible patient, may cause an exaggerated QT prolongation.1 Another reason for the variability in risk for torsade de pointes relates to genetic susceptibility for this arrhythmia. These factors control the duration of the QT interval. At least 6 separate genes, if mutated, can cause the congenital long-QT interval. In particular, the human ether-a-go-go related gene (HERG), which encodes a potassium-channel protein that regulates repolarization potassium currents, has been implicated in increasing the risk of drug-induced torsade de pointes.

A number of drugs used by physicians in the perioperative period effect the QT interval. These include the anti-arrhythmic agents, calcium-channel blockers, antibiotics, antipsychotic drugs, and antiemetic agents like droperidol and haloperidol. Any agent which results in a QT prolongation greater than 500 ms is thought to significantly escalate the possibility of developing this arrhythmia. Drugs which increases that QT interval more than 500 ms should be immediately discontinued (normal values for the QT interval are < 430 ms in males and < 450 ms in females). According to guidelines published by the European Agency for the Evaluation of Medicinal Products, drugs which induce individual changes in the QT of 30 ms are unlikely to raise concerns about arrhythmias, changes of 30-60 ms are thought to potentially increase the risk for arrhythmias, and drug-effects which raise the QT interval more than 60 ms increase concerns about arrythmogenic risk.

Oral methadone is a long acting agent which has been traditionally used to treat opioid addiction. In addition, it is being increasingly used as an important therapy for chronic pain. This agent has a long half-life and can be administered once daily. In addition to its analgesic effects due to its long-acting agonist effect on the µ-receptor, methadone is an antagonist of the N-methyl-D-aspartate (NMDA) receptor. Antagonism of the NMDA receptor may play an important role in treating acute pain and preventing the development of chronic postoperative pain. Furthermore, methadone may prevent reuptake of the neurotransmitters norepinephrine and serotonin and result in improved mood states. In chronic pain patients, methadone may be more effective in treating neuropathic pain and prevent the development of tolerance. Despite these potential advantages, patients receiving chronic methadone therapy are at increased risk of cardiac death. Methadone has been reported to be implicated in 30-40% of opioid-related deaths. Although a number of these deaths may be related to respiratory depression, others may be due to QT prolongation and torsade de pointes. Risk factors in these patients for lethal arrhythmias include dose of methadone, duration of treatment, electrolyte abnormalities, older age, female sex, cirrhosis, genetic susceptibility, and use of other drugs that prolong the QT interval. Studies have demonstrated a mean increase in the QT interval of 15 ms and 34 ms in patients on chronic methadone treatment.

Over the past decade, the use of intravenous methadone in the operating room setting has dramatically increased. An important limitation of the intravenous opioids typically used in the operating room and in the postoperative period for pain management is that the duration of effect of these agents is only 3 to 4 hours. This results in periods of effective pain relief, followed by periods of moderate-to-severe pain in the postoperative period. An alternative strategy for opioid utilization may involve the administration of a very long-acting opioid in the operating room that would provide effective analgesia for the first 24 postoperative hours (which corresponds with the period of the most severe pain after surgery). At the present time, intravenous methadone is the only long-acting opioid available to anesthesiologists. A primary advantage of methadone is its long half-life, which ranges from 25-52 hours when given intravenously in larger doses. Therefore, a single dose given at induction of anesthesia can be used in patients with moderate-to-severe to provide analgesia throughout the perioperative period. In randomized, double-blinded investigations in cardiac and orthopedic surgical patients, subjects randomized to the methadone group reported less pain, required reduced postoperative analgesic medications, and described increased satisfaction with overall pain management when compared to subjects administered a standard opioids.

No adverse events directly attributable to methadone were reported in any clinical trials using methadone in the operating room. In particular, no cardiac events, episodes of QT prolongation, or observations of torsade de pointes were reported in any studies. In addition, no case reports of adverse cardiac events related to methadone have been described in the literature. However, none of the previous studies have specifically assessed the effect of methadone on the incidence of QT prolongation or obtained postoperative EKGs. Only two previous investigations have examined the potential effects of a single dose of methadone on the QT interval. In dogs given 0.3 to 1.0 mg/kg doses of intravenous methadone, no significant effect on the QRS duration or QT interval was observed. In a post-hoc analysis of data from a randomized study examining the effect of vitamin treatment and nitrous oxide on cardiovascular events, the impact of various anesthetic agents on the QT interval was examined. EKGs were obtained before anesthesia, 30 minutes after PACU admission, and on postoperative days 1 and 2. Eighty percent of patients had significant QT prolongation in the PACU, whereas no patient had QT prolongation by postoperative day 1. Several drugs were associated with increases in the QT interval, including inhalational agents, ketorolac, antibiotics, vasoactive drugs, and methadone. Fifty-three percent of the patients administered methadone had a QT interval increase of > 30 ms. An important limitation of this investigation is that it was a post-hoc analysis of data from a study in which anesthetic care was not standardized. The data demonstrates, however, that a number of anesthetic agents increase the QT interval. In addition, the stress response to surgery has been demonstrated to increase the QT interval. Despite the frequent use of these agents in the operating room, torsade de pointes is a rare event during or immediately following surgery.

At the present time, no previous randomized trials have assessed the effect of a single dose of methadone, given at induction of anesthesia, on the QT interval as a primary endpoint. The aim of this clinical investigation is to examine the impact of a standard dose of perioperative methadone (0.2 mg/kg ideal body weight (IBW)) on the QT interval, measured with a 12-lead EKG, 30 minutes after PACU admission and on the morning of postoperative day 1. We hypothesize that patients randomized to receive methadone will not have a higher incidence of QT prolongation, when compared to patients given a dose of hydromorphone (the standard intraoperative opioid administered to patients undergoing procedures associated with moderate-to-severe postoperative pain). Secondary endpoints include levels of postoperative pain, analgesic requirements, and any opioid-related complications (level of sedation, episodes of respiratory complications)

ELIGIBILITY:
Inclusion Criteria:

* All patients presenting for elective surgical cases requiring general anesthesia and associated with moderate-to-severe postoperative pain will be eligible for enrollment.

Exclusion Criteria:

* History of arrhythmias, pacemaker, or defibrillator
* Allergy to methadone or hydromorphone
* Preoperative altered mental status
* Abnormal serum electrolyte values
* Existence of significant valvular disease or cardiac rhythm other than sinus
* Significant preoperative pain requiring treatment with opioids or recent history of opioid abuse

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2020-08-12 (Estimated); Study Completion 2020-12-23 (Estimated)

PRIMARY OUTCOMES:
QT prolongation on the EKG 30 minutes after postanesthesia care unit admission | 30 minutes after post anesthesia care unit admission
  EKGs will be obtained 30 minutes after postanesthesia care unit admission

SECONDARY OUTCOMES:
QT prolongation on the EKG on the morning of postoperative day one | 24 hours after surgery
  EKGs will be obtained on the morning of postoperative day one
Level of pain on on a 0-10 scale 30 minutes after postanesthesia care unit admission | 30 minutes after postanesthesia care unit admission
  Pain will be assessed on a 0-10 scale (0=no pain, 10 worst pain imaginable)
Level of pain on a 0-10 scale on the morning of postoperative day one | 24 hours after surgery
  Pain will be assessed on a 0-10 scale (0=no pain, 10 worst pain imaginable)

CONTACTS AND LOCATIONS:
Overall Officials: Glenn S Murphy, MD, Principal Investigator — Endeavor Health
Locations (1):
- NorthShore University HealthSystem, Evanston, Illinois, United States

IPD SHARING:
Plan to Share IPD: No